CLINICAL TRIAL: NCT03239951
Title: One-arm, Controlled, Multi-Center Prospective Study to Assess the Efficacy, Safety and Tolerability of Medi-Tate Temporary Implantable Nitinol Device (iTind) in Subjects With Acute Urinary Retention Secondary to (BPO)
Brief Title: Study to Assess the Efficacy, Safety and Tolerability of (iTind)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 outbreak and the overall low recruitment
Sponsor: Medi-Tate Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-04
Record Dates: First submitted 2017-07-25; First posted 2017-08-04 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: BPH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device (Experimental): Temporary implant (iTind)
  Interventions: Device: iTind

INTERVENTIONS:
Device: iTind — temporary implant

SUMMARY:
Subjects with AUR secondary to BPO that comply with Inclusion/Exclusion Criteria.

A total of 50 eligible subjects will be recruited into the study to receive treatment with iTind system.

Study duration will be 12 months post implantation, with follow-up extension of up to 3 years. Extension of follow up period will not require an additional ICF.

DETAILED DESCRIPTION:
Spontaneous acute urinary retention (AUR) is one of the most significant complications of long-term benign prostatic hyperplasia (BPH). In the past it has represented an immediate indication for surgery. Between 25% and 30% of men who underwent transurethral prostatectomy (TURP) had AUR as their main indication in older series and today most subjects failing to void after attempted catheter removal still undergo surgery. For this reason alone, AUR is an important and feared event from the viewpoint of the subject. The subject originally has inability to urinate, with increasing pain, and eventually a visit to the emergency room, catheterization, follow-up visits to the physicians, an attempt at catheter removal, and eventual recovery or surgery, which is both painful and time consuming.

After the acute period most men with AUR will be offered a 'trial without catheter' (TWOC) and about half will resume spontaneous voiding. Most men who fail a TWOC, experience a recurrent episode of AUR, or have moderate or severe lower urinary tract symptoms (LUTS) that are refractory to medical management will be considered for surgery.

In the older literature, the risk of recurrent AUR was cited as 56% to 64% within 1 week of the first episode and 76% to 83% in men with diagnosed BPH.

(http://www.ncbi.nlm.nih.gov/pmc/articles/PMC1476058/). Additional researches show that ten percent of men in their seventies and 30% in their eighties will have AUR within the next five years.

Benign prostatic hyperplasia is the cause for the AUR in at least 65% of men presenting with AUR.

In the below study of the natural history of BPH, the risk of AUR was 1.6% at five years for men aged 40-49 years and 10% at 70-79 years.

ELIGIBILITY:
Inclusion Criteria:

* Male with AUR secondary to BPO
* Age ≥40 years
* Acute urinary retention with at least one failed trial without catheter (TWOC) while on alpha blocker
* Ability to sign an informed consent form
* Prostate volume <80 ml
* Life expectancy >1 year.

Exclusion Criteria:

* Suspected malignant disease of the lower urinary tract including prostate or bladder cancer
* Chronic retention of urine with history of either retention volume greater than one liter or upper tract obstruction
* Known neurogenic bladder
* Immunosuppression
* Suspected urethral strictures, bladder neck contracture, Urinary bladder stones
* An obstructive or protruding median lobe of the prostate
* An active symptomatic urinary tract infection
* Enrolled in another treatment trial for any disease
* Previous pelvic irradiation or radical pelvic surgery
* Any previous prostate surgery.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Ability to void without catheter | 2 weeks
  TWOC Success Rate, defined as the proportion (%) of subjects successfully undergoing the TWOC assessment at the later of visit 3 or visit 4.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Muir, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - Firmly Park Hospital, Frimley
  - King's college, London
  - Norwich University Hospital, Norwich